CLINICAL TRIAL: NCT02243345
Title: Delayed Recompression for Decompression Sickness
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 134/13
Record Dates: First submitted 2014-09-10; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Recompression Treatment After Decompression Sickness
Keywords: decompression; recompression; delayed; late

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Delayed: Time from surfacing to recompression >=48 hours
- Early: Time from surfacing to recompression <48 hours

SUMMARY:
Decompression sickness syndrome (DCS) is caused by microbubbles forming in blood vessels or tissues during a reduction in environmental pressure (decompression). Bubbles have mechanical, embolic and biochemical effects with manifestations ranging from none to fatal. By reducing bubble volume and hastening inert gas elimination, recompression therapy with hyperbaric treatment remains the main therapy for DCS. The most common hyperbaric protocol used, is based on US Navy Treatment table 6, started as early as possible after surfacing. The outcome of hyperbaric therapy varies with reported complete resolution in 13%-63% of the patients suffering from severe DCS, and in 73%-100% of the patients with mild-moderate DCS.

The significance of time to recompression is controversial. It has been suggested that early hyperbaric treatment improves the outcome by decreasing bubble size and avoiding further tissue injury. However, in recent studies time to recompression had very little effect on clinical recovery. Moreover, the time beyond which hyperbaric treatment isn't effective has not been determined yet.

The aim of this study was to evaluate the clinical outcome of delayed hyperbaric treatment to divers who referred to tertiary care hospital hyperbaric unit, more than 48 hours after surfacing. The clinical outcome of the delayed hyperbaric treatments was compared to early treatments given at the same hyperbaric unit.

DETAILED DESCRIPTION:
From January 2000 to February 2014, 204 divers were treated for DCS in the institute of Hyperbaric Medicine, Assaf Harofeh Medical Center, Israel.

The data will be collected retrospectively from medical records and include age, sex, diving experience, maximal depth, DCS possible cause, DCS type, symptoms, time from surfacing to symptoms onset, time from surfacing to recompression, recompression table, additional treatment after the first recompression and treatment outcome.

Statistical analysis will be done using univariant analysis was performed using Spearman's correlation and Chi-Square in categoric variabales, independent t-test in numeric variables. This will be performed in SPSS v.21 software.

ELIGIBILITY:
Inclusion Criteria:

* Decompression sickness after diving
* Recompression Treatment between 2000-2014 in Assaf HaRofe medical center hyperbaric institute

Exclusion Criteria:

* Decompression sickness excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Decompression sickness patients treated with hyperbaric recompression
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Clinical outcome evaluation | 14 days after treatment
  Clinical outcome will be reviewed from the medical records. The outcome was evaluated by a hyperbaric physician within 14 days from recompression. The outcome will be scored as complete, partial or no recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Study Chair — Assaf Harofe Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel, Israel